CLINICAL TRIAL: NCT04402866
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Parallel-group, Multi-center Study of an Inhaled Pan-Janus Kinase Inhibitor, TD-0903, to Treat Symptomatic Acute Lung Injury Associated With COVID-19
Brief Title: TD-0903 for ALI Associated With COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0188; 2020-001807-18 (EudraCT Number)
Record Dates: First submitted 2020-05-22; First posted 2020-05-27 (Actual); Results first posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Acute Lung Injury (ALI) Associated With COVID-19; Lung Inflammation Associated With COVID-19
Keywords: Acute lung injury; ALI; COVID-19; Coronavirus Disease 2019; inflammatory lung conditions; Inflammatory lung disease; ARDS; SARS-CoV-2; Pneumonia
MeSH Terms: conditions — Acute Lung Injury; COVID-19; Pneumonia | interventions — nezulcitinib

STUDY DESIGN:
Intervention Model Description: Parallel group, randomized, double-blind, placebo-controlled
Who Masked: Participant, Care Provider, Investigator
Masking Description: Pharmacist & Sponsor are not blinded for Part 1. Sponsor is blinded for Part 2. Pharmacist is not blinded for Part 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Part 1: TD-0903 - MAD Dose A (Experimental): 6 out of 8 subjects per cohort will be randomized to receive TD-0903 MAD Dose A
  Interventions: Drug: TD-0903
- Part 1: TD-0903 - MAD Dose B (Experimental): 6 out of 8 subjects per cohort will be randomized to receive TD-0903 MAD Dose B
  Interventions: Drug: TD-0903
- Part 1: TD-0903 - MAD Dose C (Experimental): 6 out of 8 subjects per cohort will be randomized to receive TD-0903 MAD Dose C
  Interventions: Drug: TD-0903
- Part 1: Placebo for MAD (Experimental): 2 out of 8 subjects per cohort (up to 3 cohorts) will be randomized to receive placebo
  Interventions: Drug: Placebo
- Part 2: TD-0903 (Experimental): 99 subjects will be randomized to receive TD-0903
  Interventions: Drug: TD-0903
- Part 2: Placebo (Experimental): 99 subjects will be randomized to receive Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TD-0903 — Study Drug to be administered by inhalation
  Arms: Part 1: TD-0903 - MAD Dose A; Part 1: TD-0903 - MAD Dose B; Part 1: TD-0903 - MAD Dose C; Part 2: TD-0903
Drug: Placebo — Placebo to be administered by inhalation
  Arms: Part 1: Placebo for MAD; Part 2: Placebo

SUMMARY:
This Phase 2 study will evaluate the efficacy, safety, pharmacodynamics and pharmacokinetics of inhaled TD-0903 compared with a matching placebo in combination with standard of care (SOC) in hospitalized patients with confirmed COVID-19 associated acute lung injury and impaired oxygenation.

DETAILED DESCRIPTION:
Part 1 of the study includes up to 3 ascending dose cohorts, each comprised of 8 subjects (6 receiving TD-0903 and 2 receiving placebo).

Part 2 of the study will evaluate one dose of TD-0903 (selected based on the data from Part 1) as compared with placebo. Part 2 is targeting 198 subjects total.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent on their own prior to performing study procedures. In the U.K., subject assent or proxy consent as per local site procedures, may also be acceptable if both a clinician and second health professional attest that the subject understands the risks and potential benefits of the study and elects to proceed. Outside the U.K., written informed consent may only be obtained from the subject or legally authorized representative. In the event the subject loses capacity during the study, the subject consents to continued participation, except where this is not clinically indicated.
* Willing and able to comply with study-related procedures/assessments
* Age 18 to 80 years old
* Hospitalized (or documentation of a plan to admit to the hospital if the subject is in an emergency department) and requiring supplemental oxygen to maintain saturation > 90%
* A diagnosis of symptomatic COVID-19 defined as a positive test for SARS-CoV-2 RNA detected by RT-PCR on a sample from the upper respiratory tract (e.g., nasopharyngeal, nasal, or oropharyngeal swab) collected < 72 hours prior to randomization
* Onset of COVID-19 -related symptoms > 2 days and </= 10 days prior to hospital admission

Exclusion Criteria:

* Subjects currently receiving invasive mechanical ventilation
* Presence or suspicion of active malignancy with the exception of cancer in situ (e.g., skin cancer)
* Evidence of serious active infection other than COVID-19
* Current diagnosis of human immunodeficiency virus, hepatitis B or C
* In the opinion of the investigator, unlikely to survive for > 24 hours from enrollment
* Women who are pregnant or might be pregnant, or who are currently breast-feeding. Subjects must agree to not donate ova or sperm through 30 days after the last dose of study medication
* Presence of significant comorbidity that, in the opinion of the investigator, predisposes the subject to mortality. Such conditions might include: a. New York Heart Association class IV Heart Failure b. Hepatic dysfunction (i.e., AST or ALT >3x upper limit of normal) c. Renal dysfunction (i.e., estimated glomerular filtration rate (eGFR) < 50mL/min) or receiving renal replacement therapy
* Presence of septic shock at time of enrollment
* Hemoglobin < 80 g/L
* Evidence of neutropenia (i.e., absolute neutrophil count < 1000 cells/uL), lymphopenia (i.e., absolute lymphocyte count < 200 cells/uL) or thrombocytopenia (i.e.Platelets < 50×10^9/L)
* Hypersensitivity to TD-0903 or its components, or to other JAK inhibitors
* Treatment with anti-IL 6 (e.g., tocilizumab, sarilumab), anti-IL-6R antagonists (e.g., abatacept), JAK inhibitors (e.g., baricitinib, tofacitinib) supplemental interferon therapy, or tyrosine kinase inhibitors (e.g., erlotinib, gefinitib) in the past 30 days, or plans to receive a JAK inhibitor during the study period
* Current treatment with conventional synthetic disease-modifying anti-rheumatic drugs (DMARDs)/immunosuppressive agents including:

  1. Methotrexate, cyclosporine, mycophenolate, tacrolimus, penicillamine, or sulfasalazine within 2 weeks prior to enrollment
  2. Azathioprine or cyclophosphamide within 12 weeks prior to enrollment
  3. Monoclonal antibodies targeting B cells (e.g., rituximab) within 12 weeks prior to enrollment
  4. Tumor necrosis factor-alpha (TNFα)) inhibitors within 4 weeks prior to enrollment
* Participating in other clinical trials involving any other experimental treatment for COVID-19, except in the context of a single-arm antiviral or convalescent plasma compassionate-use protocol
* Subjects with active or incompletely treated pulmonary tuberculosis, or known history of non-tuberculosis mycobacterium over past 12 months
* Subject requires continuous oxygen supplementation for underlying cardio-respiratory history in the past 90 days
* Body Mass Index ≥40 kg/m2
* Receipt of live vaccine (i.e., live attenuated) in the 4 weeks prior to visit 1 or plans to receive a live vaccine (or live attenuated) during the study period. Note: Use of non-live (inactivated) vaccinations is allowed for all subjects
* History of venous thromboembolism (VTE), deep venous thrombosis (DVT), Pulmonary Embolism (PE) or known hypercoagulable disorder (e.g., factor V Leiden, antiphospholipid antibody syndrome, protein C or S deficiency)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2020-06-24 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2021-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (23):
- United States (12):
  - Theravance Biopharma Investigational Site, Duarte, California
  - Theravance Biopharma Investigational Site, Denver, Colorado
  - Theravance Biopharma Investigational Site, Sebring, Florida
  - Theravance Biopharma Investigational Site, Boston, Massachusetts
  - Theravance Biopharma Investigational Site, Fall River, Massachusetts
  - Theravance Biopharma Investigational Site, Kalispell, Montana
  - Theravance Biopharma Investigational Site, Glens Falls, New York
  - Theravance Biopharma, Hyde Park, New York
  - Theravance Biopharma Investigational Site, Columbus, Ohio
  - Theravance Biopharma Investigational Site, Allentown, Pennsylvania
  - Theravance Biopharma Investigational Site, Bethlehem, Pennsylvania
  - Theravance Biopharma Investigational Site, Wenatchee, Washington
- Brazil (4):
  - Theravance Biopharma Investigational Site, Bela Vista
  - Theravance Biopharma Investigational Site, Botucatu
  - Theravance Biopharma Investigational Site, Caxias do Sul
  - Theravance Biopharma Investigational Site, São José do Rio Preto
- Finland (2):
  - Theravance Biopharma Investigational Site, Helsinki
  - Theravance Biopharma Investigational Site, Turku
- Theravance Biopharma Investigational Site, Chisinau, Moldova
- Theravance Biopharma Investigational Site, Bucharest, Romania
- Ukraine (2):
  - Theravance Biopharma Investigational Site, Brovary
  - Theravance Biopharma Investigational Site, Kyiv
- Theravance Biopharma Investigational Site, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Theravance Biopharma, Inc. will not be sharing individual de-identified participant data or other relevant study documents.

REFERENCES:
- [Derived] Belperio J, Nguyen T, Lombardi DA, Bogus M, Moskalenko V, Singh D, Haumann B, Bourdet DL, Kaufman E, Pfeifer ND, Thompson CG, Woo J, Moran EJ, Saggar R. Efficacy and safety of an inhaled pan-Janus kinase inhibitor, nezulcitinib, in hospitalised patients with COVID-19: results from a phase 2 clinical trial. BMJ Open Respir Res. 2023 Jul;10(1):e001627. doi: 10.1136/bmjresp-2023-001627. PMID 37460276

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 235 participants were enrolled across 24 sites in the United States, Brazil, Finland, the Republic of Moldova, Romania, Ukraine and the United Kingdom.
Pre-assignment Details: 235 participants were enrolled and 230 participants were randomized and treated with study drug. Within each cohort in Part 1 (multiple-ascending dose design), participants were randomized 3:1, TD-0903 to placebo. During Part 2 (parallel-group design), participants were stratified by baseline age (≤ 60 versus > 60 years), and by concurrent use of antiviral medications (yes or no) at baseline. Within each stratum, participants were randomized 1:1 to receive either TD-0903 or placebo.
Groups:
- Part 1: Matching Placebo; Part 2: Matching Placebo: Matching placebo inhalation solution (1 mL) was administered once daily for up to 7 days via oral inhalation using the Aerogen Solo nebulizer system.
- Part 1: TD-0903 - 1 mg: TD-0903 inhalation solution (1 mL) was administered once daily for up to 7 days via oral inhalation using the Aerogen Solo nebulizer system at a dose of 1 mg. Participants were administered a 2 mg loading dose as the total dose on Day 1.
- Part 1: TD-0903 - 3 mg; Part 2: TD-0903 - 3 mg: TD-0903 inhalation solution (1 mL) was administered once daily for up to 7 days via oral inhalation using the Aerogen Solo nebulizer system at a dose of 3 mg. Participants were administered a 6 mg loading dose as the total dose on Day 1.
- Part 1: TD-0903 - 10 mg: TD-0903 inhalation solution (1 mL) was administered once daily for up to 7 days via oral inhalation using the Aerogen Solo nebulizer system at a dose of 10 mg.
Period: Overall Study
Arm/Group | Part 1: Matching Placebo | Part 1: TD-0903 - 1 mg | Part 1: TD-0903 - 3 mg | Part 1: TD-0903 - 10 mg | Part 2: Matching Placebo | Part 2: TD-0903 - 3 mg
Started | 6 | 6 | 7 | 6 | 104 | 106
Randomized and Treated With Study Drug | 6 | 6 | 7 | 6 | 102 | 103
Completed | 4 | 5 | 6 | 6 | 89 | 92
Not Completed | 2 | 1 | 1 | 0 | 15 | 14
Not completed — Discontinued Prior to Treatment | 0 | 0 | 0 | 0 | 2 | 3
Not completed — Adverse Event | 2 | 1 | 0 | 0 | 13 | 8
Not completed — Miscellaneous | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Part 1: Safety analysis set - all participants who received at least one dose of study drug.
  Part 2: Intent-to-Treat (ITT) analysis set - all participants who were randomized into the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Matching Placebo | Part 1: TD-0903 - 1 mg | Part 1: TD-0903 - 3 mg | Part 1: TD-0903 - 10 mg | Part 2: Matching Placebo | Part 2: TD-0903 - 3 mg | Total
Number analyzed (Participants) | 6 | 6 | 7 | 6 | 104 | 106 | 235
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 5 | 5 | 70 | 60 | 146
  >=65 years | 3 | 3 | 2 | 1 | 34 | 46 | 89
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 3 | 1 | 41 | 41 | 90
  Male | 3 | 5 | 4 | 5 | 63 | 65 | 145
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 10 | 14 | 24
  Not Hispanic or Latino | 6 | 6 | 7 | 6 | 90 | 89 | 204
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 4 | 3 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0 | 0 | 2 | 2
  White | 5 | 6 | 7 | 6 | 102 | 104 | 230
  More than one race | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Other | 0 | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Part 2: Number of Respiratory Failure-free Days (RFDs) From Randomization to Day 28
Description: An RFD was defined as a day that a participant was alive and did not require the use of any respiratory support (invasive mechanical ventilation, non-invasive positive pressure ventilation, high-flow oxygen devices, or oxygen supplementation) from randomization through Day 28. The number of RFDs was 0 for participants who used respiratory support for 28 days or longer or for participants who died on or before Day 28.
  A clinical status score of ≤ 4 on a given day was equivalent to an RFD. The clinical status categories and associated scores ranged from 1-8 where a higher score represented a worse outcome. A clinical status score of 4 was defined as a participant who was hospitalized, not requiring supplemental oxygen, but requiring ongoing medical care (whether or not related to COVID-19).
Time Frame: Randomization to Day 28
Population: ITT analysis set (Part 2) - all participants with analyzable data who were randomized into the study.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Part 2: Matching Placebo | Part 2: TD-0903 - 3 mg
Number analyzed (Participants) | 102 | 100
days | 21.0 [15.0 to 23.0] | 21.0 [17.5 to 23.0]
Statistical Analysis 1: Comparison: Part 2: Matching Placebo vs Part 2: TD-0903 - 3 mg; Since this was a Phase 2 study, it was not powered for any of the secondary endpoints; Test type: Other; p = 0.6137, Van Elteren test; Common Odds Ratio = 1.142, 95% CI 2-sided [0.706 to 1.846] — Common Odds Ratio (TD-0903 vs. placebo) and corresponding 95% Wald confidence interval (CI) were obtained from the proportional odds regression model of RFD adjusting for baseline age strata (≤ 60 years vs. > 60 years)

2. Secondary Outcome: Part 2: Change From Baseline in SaO2/FiO2 Ratio on Day 7
Description: SaO2/FiO2 ratio was calculated as SaO2 divided by FiO2.
Time Frame: Baseline and Day 7
Population: ITT analysis set (Part 2) - all participants with analyzable data who were randomized into the study.
Measure: Least Squares Mean (Standard Error); unit: ratio measure
Arm/Group | Part 2: Matching Placebo | Part 2: TD-0903 - 3 mg
Number analyzed (Participants) | 86 | 90
ratio measure | 88.97 (7.769) | 88.46 (7.654)
Statistical Analysis 1: Comparison: Part 2: Matching Placebo vs Part 2: TD-0903 - 3 mg; Part 2: TD-0903 - Parallel-Group 3 mg versus Part 2: Matching Placebo - Parallel-Group; Test type: Other — Since this was a Phase 2 study, it was not powered for any of the secondary endpoints; p = 0.962, Mixed model repeated measures model; LS mean difference = -0.51, 95% CI 2-sided [-21.95 to 20.92]

3. Secondary Outcome: Part 2: Number of Participants in Each Category of the 8-point Ordinal Clinical Status Scale on Days 7, 14, 21, and 28
Description: The clinical status categories and associated scores ranged from 1-8 where a higher score represented a worse outcome. The scale was as follows:
  * Score 1: Not hospitalized, no limitations on activities
  * Score 2: Not hospitalized, but with limitations on activities and/or requiring home oxygen
  * Score 3: Hospitalized, not requiring supplemental oxygen, and no longer requiring ongoing medical care
  * Score 4: Hospitalized, not requiring supplemental oxygen, but requiring ongoing medical care (whether or not related to COVID-19)
  * Score 5: Hospitalized, requiring supplemental oxygen
  * Score 6: Hospitalized, on non-invasive ventilation or high-flow oxygen devices
  * Score 7: Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation
  * Score 8: Death
Time Frame: Days 7, 14, 21 and 28
Population: ITT analysis set (Part 2) - all participants with analyzable data who were randomized into the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Matching Placebo | Part 2: TD-0903 - 3 mg
Number analyzed (Participants) | 102 | 100
Participants
  Day 7: number analyzed (Participants) | 102 | 99
  Day 7: Score 1 | 6 | 8
  Day 7: Score 2 | 12 | 9
  Day 7: Score 3 | 1 | 1
  Day 7: Score 4 | 25 | 23
  Day 7: Score 5 | 42 | 48
  Day 7: Score 6 | 7 | 7
  Day 7: Score 7 | 7 | 2
  Day 7: Score 8 | 2 | 1
  Day 14: number analyzed (Participants) | 102 | 99
  Day 14: Score 1 | 57 | 52
  Day 14: Score 2 | 6 | 11
  Day 14: Score 3 | 2 | 7
  Day 14: Score 4 | 14 | 13
  Day 14: Score 5 | 10 | 7
  Day 14: Score 6 | 1 | 2
  Day 14: Score 7 | 6 | 5
  Day 14: Score 8 | 6 | 2
  Day 21: number analyzed (Participants) | 102 | 99
  Day 21: Score 1 | 72 | 72
  Day 21: Score 2 | 4 | 9
  Day 21: Score 3 | 4 | 6
  Day 21: Score 4 | 4 | 0
  Day 21: Score 5 | 3 | 4
  Day 21: Score 6 | 1 | 0
  Day 21: Score 7 | 2 | 3
  Day 21: Score 8 | 12 | 5
  Day 28: Score 1 | 79 | 78
  Day 28: Score 2 | 5 | 11
  Day 28: Score 3 | 0 | 1
  Day 28: Score 4 | 1 | 1
  Day 28: Score 5 | 3 | 1
  Day 28: Score 6 | 0 | 0
  Day 28: Score 7 | 1 | 2
  Day 28: Score 8 | 13 | 6
Statistical Analysis 1: Comparison: Part 2: Matching Placebo vs Part 2: TD-0903 - 3 mg; Part 2: TD-0903 - Parallel-Group 3 mg versus Part 2: Matching Placebo - Parallel-Group on Day 7; Test type: Other — Since this was a Phase 2 study, it was not powered for any of the secondary endpoints; p = 0.5918, Van Elteren test; Odds Ratio (OR) = 1.153, 95% CI 2-sided [0.692 to 1.922] — Between-group comparisons analyzed using a proportional odds model adjusting for baseline age strata (≤ 60 years vs. > 60 years)
Statistical Analysis 2: Comparison: Part 2: Matching Placebo vs Part 2: TD-0903 - 3 mg; Part 2: TD-0903 - Parallel-Group 3 mg versus Part 2: Matching Placebo - Parallel-Group on Day 14; Test type: Other — Since this was a Phase 2 study, it was not powered for any of the secondary endpoints; p = 0.6978, Van Elteren test; Odds Ratio (OR) = 1.105, 95% CI 2-sided [0.651 to 1.878]; Between-group comparisons analyzed using a proportional odds model adjusting for baseline age strata (≤ 60 years vs. > 60 years)
Statistical Analysis 3: Comparison: Part 2: Matching Placebo vs Part 2: TD-0903 - 3 mg; Part 2: TD-0903 - Parallel-Group 3 mg versus Part 2: Matching Placebo - Parallel-Group on Day 21; Test type: Other — Since this was a Phase 2 study, it was not powered for any of the secondary endpoints; p = 0.3990, Van Elteren test; Odds Ratio (OR) = 1.295, 95% CI 2-sided [0.702 to 2.388]; [other analysis details as in outcome 3, analysis 2]
Statistical Analysis 4: Comparison: Part 2: Matching Placebo vs Part 2: TD-0903 - 3 mg; Part 2: TD-0903 - Parallel-Group 3 mg versus Part 2: Matching Placebo - Parallel-Group on Day 28; Test type: Other — Since this was a Phase 2 study, it was not powered for any of the secondary endpoints; p = 0.6445, Van Elteren test; Odds Ratio (OR) = 1.180, 95% CI 2-sided [0.605 to 2.299] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Part 2: Number of Participants Alive and Respiratory Failure-free on Day 28
Description: Defined as participants who were alive and did not require the use of any respiratory support (invasive mechanical ventilation, non-invasive positive pressure ventilation, high-flow oxygen devices, or oxygen supplementation) on Day 28.
Time Frame: Day 28
Population: ITT analysis set (Part 2) - all participants with analyzable data who were randomized into the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Matching Placebo | Part 2: TD-0903 - 3 mg
Number analyzed (Participants) | 104 | 106
Participants | 85 | 92
Statistical Analysis 1: Comparison: Part 2: Matching Placebo vs Part 2: TD-0903 - 3 mg; Part 2: TD-0903 - Parallel-Group 3 mg versus Part 2: Matching Placebo - Parallel-Group; Test type: Other — Since this was a Phase 2 study, it was not powered for any of the secondary endpoints; p = 0.3005, Cochran-Mantel-Haenszel chi-square test — The p-value was calculated using the Cochran-Mantel-Haenszel chi-square test stratified by baseline age group (≤ 60 years vs. > 60 years); Risk Difference (RD) = 5.06, 95% CI 2-sided [-4.50 to 14.63]

ADVERSE EVENTS:
Time Frame: Day 1 to Day 28
Description: Safety analysis set - all participants who received at least one dose of study drug.
Groups:
- Part 1: TD-0903 - 1 mg: TD-0903 inhalation solution (1 mL) was administered once daily for up to 7 days via oral inhalation using the Aerogen Solo nebulizer system at a dose of 1 mg.
- Part 1: TD-0903 - 3 mg: TD-0903 inhalation solution (1 mL) was administered once daily for up to 7 days via oral inhalation using the Aerogen Solo nebulizer system at a dose of 3 mg.
- Part 2: TD-0903 - 3 mg: TD-0903 inhalation solution (1 mL) was administered once daily for up to 7 days via oral inhalation using the Aerogen Solo nebulizer system. Participants were administered the recommended dose of 3 mg based on the data from Part 1.
Arm/Group | Part 1: Matching Placebo | Part 1: TD-0903 - 1 mg | Part 1: TD-0903 - 3 mg | Part 1: TD-0903 - 10 mg | Part 2: Matching Placebo | Part 2: TD-0903 - 3 mg
All-Cause Mortality (participants affected / at risk) | 2/6 | 1/6 | 0/7 | 0/6 | 13/102 | 6/103
Serious Adverse Events (participants affected / at risk) | 3/6 | 1/6 | 1/7 | 0/6 | 16/102 | 10/103
Other Adverse Events (participants affected / at risk) | 6/6 | 4/6 | 1/7 | 5/6 | 18/102 | 15/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Matching Placebo (N=6) | Part 1: TD-0903 - 1 mg (N=6) | Part 1: TD-0903 - 3 mg (N=7) | Part 1: TD-0903 - 10 mg (N=6) | Part 2: Matching Placebo (N=102) | Part 2: TD-0903 - 3 mg (N=103)
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 3
Multiple organ dysfunction syndrome (General disorders) | 1 | 1 | 0 | 0 | 1 | 3
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 3 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 3 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Shock (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 4 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 5 | 3
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Sudden death (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Systemic bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Matching Placebo (N=6) | Part 1: TD-0903 - 1 mg (N=6) | Part 1: TD-0903 - 3 mg (N=7) | Part 1: TD-0903 - 10 mg (N=6) | Part 2: Matching Placebo (N=102) | Part 2: TD-0903 - 3 mg (N=103)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 1 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 1
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1
Depressed mood (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 2 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Vascular device infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 2 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 4
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 7 | 3
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 6 | 5
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/66/NCT04402866/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-22): https://cdn.clinicaltrials.gov/large-docs/66/NCT04402866/SAP_001.pdf